CLINICAL TRIAL: NCT06108440
Title: Comparative Effects of Action Observation and Motor Imagery Training on Upper Limb Function in Chronic Stroke Patients
Brief Title: Comparative Effects of Action Observation and Motor Imagery on Upper Limb in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0232
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Upper Extremity Paresis; Motor Activity
Keywords: Stroke; Upper Extremity Paresis; Motor Activity
MeSH Terms: conditions — Stroke; Paresis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be divided into Group A (n = 20) and Group B (n = 20) using a randomization through computer generated numbers program. Patients in Group A will receive action observation training with conventional treatment. All participants will undergo the training for 25 minutes per session, 5 days per week for 8 weeks. Patients in Group B will receive motor imagery with conventional treatment. All participants will receive interventions for twenty-five minutes per session, five times a week, for eight weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- action observation training group (Experimental): Patients in Group A will receive action observation training with conventional treatment.
  Interventions: Other: action observation training
- motor imagery training group (Active Comparator): Patients in Group B will receive motor imagery with conventional treatment.
  Interventions: Other: motor imagery training

INTERVENTIONS:
Other: action observation training — Patients in Group A will receive action observation training with conventional treatment. All participants will undergo the training for 25 minutes per session, 5 days per week for 8 weeks.
  Arms: action observation training group
Other: motor imagery training — Patients in Group B will receive motor imagery with conventional treatment. All participants will receive interventions for twenty-five minutes per session, five times a week, for eight weeks.
  Arms: motor imagery training group

SUMMARY:
To Compare effects of action observation and motor imagery training on upper limb function in chronic stroke patients.

DETAILED DESCRIPTION:
The study is Randomized controlled trial. The study will be conducted on 44 stroke patients. The study will be conducted in Civil Hospital Shujaabad and Riphah rehabilitation centre Lahore. Patients will be divided into Group A (n = 20) and Group B (n = 20) using a randomization through computer generated numbers program. Patients in Group A will receive action observation training with conventional treatment. All participants will undergo the training for 25 minutes per session, 5 days per week for 8 weeks. Patients in Group B will receive motor imagery with conventional treatment. All participants will receive interventions for twenty-five minutes per session, five times a week, for eight weeks. For the pre- and post-evaluation of all participants, Fugl-Meyer Assessment Upper Extremity (FMA UE) and Wolf Motor Function Test (WMFT) will be used. Data will be analyzed by using SPSS (Statistical package for Social Sciences) 25 version.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic stroke by a neurologist
* 03 months post stroke
* Score 1+ on modified ashworth scale
* Having a score of 24 or higher in the Mini-Mental State Examination

Exclusion Criteria:

* Patient with neurological condition other than stroke e.g. Parkinson's or multiple sclerosis
* Presence of an attached artificial pacemaker
* Presence of a metal implant in the brain
* Presence of visual impairment
* Presence of unilateral neglect in Line bisection test (25)
* Use of antipsychotic drugs

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity (FMA UE): | 6 months
  Fugl-Meyer Assessment Upper Extremity (FMA UE):
  FMA UE is a detailed evaluation tool that quantitatively measures motor function, balance, sensation, joint range of motion, and pain in stroke hemiplegic patients
Wolf Motor Function Test (WMFT): | 6 months
  Wolf Motor Function Test (WMFT):
  The Wolf motor function test is a tool to evaluate upper extremity motor function in hemiplegic patients. It has 17 tasks with a score range from 0-5. The inter-rater reliability of the function score is 0.88 and the inter-rated reliability of performance time is 0.97

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demartino AM, Rodrigues LC, Gomes RP, Michaelsen SM. Hand function and type of grasp used by chronic stroke individuals in actual environment. Top Stroke Rehabil. 2019 May;26(4):247-254. doi: 10.1080/10749357.2019.1591037. Epub 2019 Mar 23. PMID 30907287
- [Background] Veldema J, Nowak DA, Gharabaghi A. Resting motor threshold in the course of hand motor recovery after stroke: a systematic review. J Neuroeng Rehabil. 2021 Nov 3;18(1):158. doi: 10.1186/s12984-021-00947-8. PMID 34732203
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218
- [Background] Serlin Y, Shelef I, Knyazer B, Friedman A. Anatomy and physiology of the blood-brain barrier. Semin Cell Dev Biol. 2015 Feb;38:2-6. doi: 10.1016/j.semcdb.2015.01.002. Epub 2015 Feb 11. PMID 25681530